CLINICAL TRIAL: NCT01140412
Title: Open-Label, Fixed-Sequence, Crossover Study To Estimate The Pharmacokinetic Interaction Between Multiple Dose Maraviroc And Fosamprenavir/Ritonavir In Healthy Subjects
Brief Title: Pharmacokinetic Interaction Between Maraviroc And Fosamprenavir/Ritonavir In Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial prematurely terminated on November 1, 2010, due to healthy volunteer participants experiencing non-serious fosamprenavir-related skin rash.
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4001099
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: maraviroc; fosamprenavir; drug interaction; pharmacokinetics; HIV; AIDS; CCR5; protease inhibitor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Twice daily regimen
  Interventions: Drug: Maraviroc; Drug: Fosamprenavir/ritonavir; Drug: Maraviroc + Fosamprenavir/ritonavir
- Cohort 2 (Experimental): Once daily regimen
  Interventions: Drug: Maraviroc; Drug: Fosamprenavir/ritonavir; Drug: Maraviroc + Fosamprenavir/ritonavir

INTERVENTIONS:
Drug: Maraviroc — maraviroc 300 mg BID x 5 days
  Other Names: Selzentry, Celsentri
  Arms: Cohort 1
Drug: Fosamprenavir/ritonavir — fosamprenavir/ritonavir 700/100 mg BID x 10 days
  Arms: Cohort 1
Drug: Maraviroc + Fosamprenavir/ritonavir — maraviroc 300 mg BID + fosamprenavir/ritonavir 700/100 mg BID x 10 days
  Arms: Cohort 1
Drug: Maraviroc — maraviroc 300 mg QD x 5 days
  Other Names: Selzentry, Celsentri
  Arms: Cohort 2
Drug: Fosamprenavir/ritonavir — fosamprenavir/ritonavir 1400/100 mg QD x 10 days
  Arms: Cohort 2
Drug: Maraviroc + Fosamprenavir/ritonavir — maraviroc 300 mg QD + fosamprenavir/ritonavir 1400/100 mg QD x 10 days
  Arms: Cohort 2

SUMMARY:
This is will be an open-label, fixed-sequence, multiple dose crossover study in 2 cohorts of 14 healthy male and/or female subjects, to estimate the effect of maraviroc on the pharmacokinetics of amprenavir and ritonavir and fosamprenavir/ritonavir on the pharmacokinetics of maraviroc.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.
* Total body weight >45 kg (99 lbs).

Exclusion Criteria:

* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Known hypersensitivity or history of allergy to sulfonamides.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maraviroc plasma pharmacokinetic parameters: AUCτ, Cmax, and Cτ on Period 1, Day 5 and Period 2, Day 20 | 25 days
Amprenavir and ritonavir plasma pharmacokinetic parameters: AUCτ, Cmax, and Cτ on Period 2, Day 10 and Period 2, Day 20 | 25 days

SECONDARY OUTCOMES:
Maraviroc plasma pharmacokinetic parameter: Tmax on Period 1, Day 5 and Period 2, Day 20. | 25 days
Amprenavir and ritonavir plasma pharmacokinetic parameter: Tmax, on Period 2, Day 10 and Period 2, Day 20. | 25 days
Safety and toleration assessed by spontaneous reporting of adverse events, vital signs, 12-lead ECG and laboratory safety assessments. | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001099&StudyName=Pharmacokinetic%20Interaction%20Between%20Maraviroc%20And%20Fosamprenavir/Ritonavir%20In%20Healthy%20Subjects%20